CLINICAL TRIAL: NCT06046833
Title: Glucose Metrics Using Freestyle Libre 3 Real-Time Continuous Glucose Monitor (rtCGM) in Patients With Gastroparesis in Type 1 or Type 2 Diabetes: Investigator Initiated Pilot Study
Brief Title: Continuous Glucose Metrics in Patients With Gastroparesis in Type 1 or Type 2 Diabetes
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Samita Garg (Other)
Responsible Party: Sponsor-Investigator, Samita Garg, Principal Investigator, The Cleveland Clinic
Organization: The Cleveland Clinic (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: 23-594
Record Dates: First submitted 2023-09-06; First posted 2023-09-21 (Actual); Last update posted 2025-04-25 (Actual); Status verified 2025-04

CONDITIONS: Diabetes Mellitus, Type 2; Diabetes Mellitus, Type 1; Gastroparesis With Diabetes Mellitus
Keywords: Gastroparesis; Diabetes; Continuous Glucose Monitor
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes Mellitus, Type 1; Gastroparesis; Diabetes Mellitus

STUDY DESIGN:
Intervention Model Description: Same intervention for two cohorts
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Patients with type 1 or type 2 diabetes and gastroparesis (Experimental): Both groups will have the same intervention.
  * FreeStyle Libre 3 sensor for Continuous Glucose Monitoring.
  * Balanced nutritional drink (Boost plus 8 ounces/237 mL) for a standardized meal challenge.
  Interventions: Device: FreeStyle Libre 3 continuous glucose monitoring sensor; Other: Nutritional drink
- Patients with type 1 or type 2 diabetes without gastroparesis (Active Comparator): Both groups will have the same intervention.
  * FreeStyle Libre 3 sensor for Continuous Glucose Monitoring.
  * Balanced nutritional drink (Boost plus 8 ounces/237 mL) for a standardized meal challenge
  Interventions: Device: FreeStyle Libre 3 continuous glucose monitoring sensor; Other: Nutritional drink

INTERVENTIONS:
Device: FreeStyle Libre 3 continuous glucose monitoring sensor — The Freestyle Libre 3 sensor is a small real-time continuous glucose monitor device that measures glucose levels every minute
  Other Names: FreeStyle Libre 3 system
Other: Nutritional drink — Balanced nutritional drink (Boost plus 8 ounces/237 mL)
  Other Names: Boost plus

SUMMARY:
A pilot study to evaluate and compare glucose metrics using a real-time continuous glucose monitor (FreeStyle Libre 3 sensor) between patients with diabetes and gastroparesis and those with diabetes without gastroparesis.

DETAILED DESCRIPTION:
Investigators will analyze and compare various Glucose Metrics (GM) derived from a Continuous Glucose Monitor (CGM) between individuals with diabetes and gastroparesis and those with diabetes without gastroparesis over a period of 28 days and during two standardized meal challenge visits. Furthermore, the investigators aim to assess whether there is an association between gastroparesis and GM parameters.

The objective is to propose a new tool (Diabetic Gastroparesis Index or Score) to assess for early gastroparesis in patients with diabetes using the identified and analyzed GM. This may help patients and providers to recognize gastroparesis early and facilitate necessary medical interventions.

Hyperglycemia and hypoglycemia episodes will be monitored throughout the study for both groups and their association with GM and gastroparesis will be evaluated.

The Gastroparesis Cardinal Symptom Index (GCSI) and the Gastrointestinal Quality of Life Index (GIQLI) questionnaires will be performed to assess the association of gastroparesis symptoms with GM.

ELIGIBILITY:
Inclusion Criteria:

* Over the age of 18 years.
* Hemoglobin A1c ≤11% within the last 6 months.
* Patients with diagnosis of type 1 Diabetes or type 2 Diabetes for at least one year.
* Normal thyroid-stimulating hormone (TSH) within the last year.
* No episodes of diabetic ketoacidosis (DKA), Hyperosmolar Hyperglycemic Status (HHS), or hypoglycemia in the past 2 weeks requiring ER visit or hospitalization.
* Symptoms of gastroparesis have been present for at least the past 3 months, in patients with gastroparesis.
* In patients with gastroparesis, documented delayed gastric emptying on scintigraphy and/or wireless motility capsule (Smart Pill) as defined by greater than 10% retention at 4 hours or greater than 4-hour gastric transit time (GTT) in the past five years.
* Patients using a Smartphone (iPhone or Android) compatible with LibreView App.

Exclusion Criteria:

* Hemoglobin A1c of >11% at enrollment.
* Advanced chronic kidney disease (serum creatinine of >2 mg/dL or estimated glomerular filtration rate (eGFR) <30mL/min/1.73m² using Chronic Kidney Disease Epidemiology Collaboration (CKD-EPI) formula).
* Advanced and significant cardiovascular disease or unstable angina.
* Advanced liver disease that may affect glucose profiles.
* Post-transplant patients.
* History of gastric surgery.
* Patients with symptoms secondary to celiac disease (e.g. diarrhea, nausea, vomiting, abdominal pain) at the time of the enrollment.
* Pregnancy or women of reproductive age group not taking adequate precautions for pregnancy for 28 days.
* Patients on steroids or immunomodulators or chemoradiation that might affect glucose profiles.
* Patients on opiates or glucagon-like peptide-1 (GLP-1) agonists (Ozempic, Wegovy, Mounjaro, Trulicity). If previously taking these medications, patients can be enrolled after 2 weeks of the last dose.
* Patient on recreational or illicit drugs (i.e., marijuana, opiates, cocaine, etc.).
* Patients on motility medications such as Reglan (Metoclopramide), Motegrity (Prucalopride), Cisapride, Domperidone, Erythromycin. If previously taking any of these medications, patients can be enrolled after 1 week of the last dose.
* Clinically significant abnormalities on upper GI endoscopy.
* Presence of imaging evidence of gastric or intestinal obstruction.
* Patient previously participated in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2024-01-08 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Time-in-Range (TIR) | 28 days of monitoring
  Percentage of time spent per day (and estimated actual amount of time in hours or minutes per day) in target glucose range 70-180 mg/dL.
Time-in-Tight Range (TITR) | 28 days of monitoring
  Percentage of time spent per day (and estimated actual amount of time in hours or minutes per day) in target glucose range 70-140 mg/dL.
Time Below Range (TBR) | 28 days of monitoring
  Percentage of time spent per day (and estimated actual amount of time in hours or minutes per day) with glucose <70 mg/dL (including readings <54 mg/dL)
Time Above Range (TAR) | 28 days of monitoring
  Percentage of time spent per day (and estimated actual amount of time in hours or minutes per day) with >180 mg/dL (including readings >250 mg/dL).
Metrics of Glucose Variability | 28 days of monitoring
  * Standard Deviation (SD)
  * Coefficient of Variation (CV)
  * Glucose Management Indicator (GMI)
  * Mean Amplitude of Glucose Excursion (MAGE)
  * Mean Of Daily Differences (MODD)
  * Mean Indices of Meal Excursion (MIME)
  * Continuous overall net glycemic action (CONGA)
  * Low Blood Glucose Index (LBGI)
  * High Blood Glucose Index (HBGI)

SECONDARY OUTCOMES:
Hyperglycemia episodes | 28 days of monitoring
  At least 15 minutes or longer of Time-Above Range (TAR) 181-250 mg/dL (Level 1 hyperglycemia) and >250 mg/dl (Level 2 hyperglycemia)
Hypoglycemia episodes | 28 days of monitoring
  At least 15 minutes or longer of Time-Below-Range (TBR) 54-69 mg/dL (Level 1 hypoglycemia) or <54 mg/dL (Level 2 hypoglycemia)

OTHER OUTCOMES:
GCSI questionnaire | Visit 2 - Day 5 (-3/+6 days), and Visit 4 - Day 25 (-7/+3 days)
  9 symptoms item questionnaire with a 6-point Likert-type response scale, ranging from 0 (none) to 5 (very severe). Total scores are in the range of 0-5, with higher scores reflecting greater symptom severity.
GIQLI questionnaire | Visit 2 - Day 5 (-3/+6 days), and Visit 4 - Day 25 (-7/+3 days)
  36-item questionnaire based on a 0-4 Likert-type scale, ranging from 0 (least desirable option) to 4 (most desirable option). Total scores range from 0 to 144, with higher scores indicating a better quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: Samita Garg, MD, Principal Investigator — The Cleveland Clinic
Locations (1):
- Cleveland Clinic Foundation, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: No